CLINICAL TRIAL: NCT06445387
Title: The Effect of Virtual Reality Glasses and Ice Applıcatıon on the Level of Pain During Femoral Sheath Removal in Patients Undergoing Percutaneous Coronary Intervenion
Brief Title: Pain During Femoral Sheath Removal in Patients Undergoing Percutaneous Coronary Intervenion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AU-SBE-ASoylu-03
Record Dates: First submitted 2024-05-16; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Percutaneous Coronary Intervention; Virtual Reality; Nursing Caries; Cryotherapy; Pain Management
Keywords: Percutaneous Coronary Intervention; Virtual Reality; Pain Management; Nursing; Ice Application
MeSH Terms: conditions — Agnosia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled, single-blind, experimental study. Participants were assigned to three groups: intervention (virtual reality group and ice group) and control group.
Who Masked: Outcomes Assessor
Masking Description: It is a randomized controlled, single-blind, experimental study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Glasses Gruop (Experimental): The procedure was tested for five minutes, one hour before application, to evaluate the patients' compliance and to detect any possible problems after wearing the glasses. In patients who did not experience any problems after the test, glasses were put on the patient just before the femoral sheath and remained on for 20 minutes.
  Interventions: Other: Virtual Reality Glasses
- Ice Application Group (Experimental): Before taking the femoral sheath, the researcher applied cold to the area where the femoral sheath was located with an ice pack for 20 minutes. A femoral sheath was performed immediately after the ice bag was removed.
  Interventions: Other: Ice Application Group
- Control Group (Other): The general procedure of the clinic was applied to the control group. Femoral sheath was removed without any invasive procedure.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Virtual Reality Glasses — Preparation Stage of Virtual Glasses: A 20-minute video consisting of nature scenes shot with a 360-degree camera was selected by the researchers from YouTube. Permission was obtained from the person who created the video.
  For the selection of music, both the music that is good for diseases were examined in the literature and an expert opinion was taken from a faculty member (Phd, assistant professor) working at the Faculty of Music and Fine Arts of a university. The music used in the video was created with works selected from the Hüseyni maqam.
  Other Names: Experimental
  Arms: Virtual Reality Glasses Gruop
Other: Ice Application Group — Features of the ice and ice bag used for patients in ice application; Ice cubes with dimensions of 9.5 x 26 x 3.5 cm were used. The ice bag is made of cotton and polyester coated fabric and is easily bendable. In this way, the ice bag was ensured to fit properly to the patient's femoral region. It is reusable and heat insulated. The procedure was carried out by following the cold application step protocol created by the researchers using the literature.
  Other Names: Experimental
  Arms: Ice Application Group
Other: Control Group — They continued to receive their routine treatment and care. No changes were made in their routine treatment and care.
  Other Names: Control
  Arms: Control Group

SUMMARY:
It is to examine the effect of virtual reality and ice application on the pain level due to femoral sheath extraction.

DETAILED DESCRIPTION:
After obtaining the necessary permissions for the research, the patients who were followed up in the hemodialysis unit of X,Y, Z Hospitals were randomly divided into three groups (virtual reality glasses application, ice application and control group).

Randomization: Since the number of male and female patients was wanted to be kept equal, simple randomization would not be possible, so the stratified randomization method was used.

Patients were assigned to groups in equal numbers according to their femoral sheath sizes. In our clinic, size 6 and 7 femoral sheaths are applied to male patients, and number 6 femoral sheaths are applied to female patients. Male patients were assigned to equal groups according to femoral sheath size 6 and 7.

Since PCI is not performed in our clinic on weekends except for emergencies, data were collected during working hours during a five-day weekday period.

The pain level of the patients was evaluated using a numerical rating scale;

* before the femoral sheath extraction (PAS1),
* during the femoral sheathing (SDQ2),
* immediately after the femoral sheathing (SDQ3),
* 30 minutes after the femoral sheathing (SDQ4) and
* 1 hour after the femoral sheathing (SDQ4). SDÖ5) was evaluated and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Intervention in the femoral region,
* Femoral sheath size is 6-7 fr,
* Presence of only one sheath in the femoral region,
* No analgesics were administered before femoral sheath removal,
* Absence of serious bleeding and major hematoma in the femoral region,
* Being over 18 years of age,
* No communication problems,
* Having a place and time orientation,
* No dizziness,
* Not having any psychiatric disease,
* No visual, auditory or mental problems,
* No previously identified cold allergy,
* Being willing and willing to participate in the study,

Exclusion Criteria:

* Serious bleeding and major hematoma development in the femoral region,
* Not applying intracoronary stent or coronary angioplasty after coronary angiography,
* Vital signs are abnormal enough to prevent intervention,
* Having visual, auditory and mental disabilities,
* Having a communication problem,
* Not being willing and able to participate in the study,
* It is defined as wanting to withdraw from the study at any stage of the study or being excluded from the study by the researcher.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — There were equal numbers of men and women in all three groups
Enrollment: 108 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Pain Scores: Numerical rating scale | "through study completion, an average of 1 year".
  The Numeric Rating Scale is a pain screening tool, commonly used to assess pain severity at that moment in time using a min:0-max:10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable" (10). This scale is a valid and reliable scale developed to determine the pain level of patients. The numerical rating scale simplifies the description of the pain level by the patient and makes it easier for the monitoring nurse to record the patient's pain rating. That the pain increases as the score increases, and then the patient verbally tells the numerical value of the pain intensity he/she feels. Pain score was measured before femoral sheath removal (time 1), and, during femoral sheath removal (2nd time),and, immediately after femoral sheath removal (3rd time), and 30 minutes after femoral sheath removal (4th time), and1 hour after femoral sheath removal (5th time).

SECONDARY OUTCOMES:
Physiological parameter | "through study completion, an average of 1 year".
  Vital parameters (Pulse rate measured in minutes) of the patients were evaluated
  Pulse rate was measured before femoral sheath removal (time 1) Pulse rate was measured during femoral sheath removal (2nd time) Pulse rate was measured immediately after femoral sheath removal (3rd time) Pulse rate was measured 30 minutes after femoral sheath removal (4th time) Pulse rate was measured 1 hour after femoral sheath removal (5th time
Physiological parameter | "through study completion, an average of 1 year".
  Vital parameters (respiration-rate measured in minutes) of the patients were evaluated.
  Respiration rate was measured before femoral sheath removal (time 1) Respiration rate was measured during femoral sheath removal (2nd time) Respiration rate was measured immediately after femoral sheath removal (3rd time) Respiration rate was measured 30 minutes after femoral sheath removal (4th time) Respiration rate was measured 1 hour after femoral sheath removal (5th time)
Physiological parameter | "through study completion, an average of 1 year".
  Vital parameters (blood pressure-measured in mmHg) of the patients were evaluated
  Blood pressure was measured before femoral sheath removal (time 1) Blood pressure was measured during femoral sheath removal (2nd time) Blood pressure was measured immediately after femoral sheath removal (3rd time) Blood pressure was measured 30 minutes after femoral sheath removal (4th time) Blood pressure was measured 1 hour after femoral sheath removal (5th time)
Physiological parameter | "through study completion, an average of 1 year".
  Vital parameters (body temperature measured in degrees Centigrant) of the patients were evaluated
  Body temperature was measured before femoral sheath removal (time 1) Body temperature was measured during femoral sheath removal (2nd time) Body temperature was measured immediately after femoral sheath removal (3rd time) Body temperature was measured 30 minutes after femoral sheath removal (4th time) Body temperature was measured 1 hour after femoral sheath removal (5th time)

OTHER OUTCOMES:
Questionnaire | "through study completion, an average of 1 year".
  The patients' opinions regarding the application of ice and virtual reality glasses were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Eylem Topbaş, Phd, Study Director — Amasya University Faculty of Health Science; Gökhan KESKİN, Phd, Study Director — Amasya University Faculty of Medical Science; Aycan SOYLU, Msc, Principal Investigator — Amasya University Instutue of Health Science
Locations (1):
- Amasya University İnstitute of Health Sciences, Amasya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
starting in December 2025
  Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR)

REFERENCES:
- [Result] Wang HL, Keck JF. Foot and hand massage as an intervention for postoperative pain. Pain Manag Nurs. 2004 Jun;5(2):59-65. doi: 10.1016/j.pmn.2004.01.002. PMID 15297952
- [Result] Paice JA, Cohen FL. Validity of a verbally administered numeric rating scale to measure cancer pain intensity. Cancer Nurs. 1997 Apr;20(2):88-93. doi: 10.1097/00002820-199704000-00002. PMID 9145556